CLINICAL TRIAL: NCT05959694
Title: A Phase Ib/II Clinical Trial on the Safety and Efficacy of TQB3909 Tablets in Patients With Recurrent or Refractory CLL/SLL.
Brief Title: A Clinical Trial on the Safety and Efficacy of TQB3909 Tablets in Patients With Recurrent or Refractory Chronic Lymphocytic Leukemia (CLL) /Small Lymphocytic Lymphoma (SLL) .
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-Ib/II-02
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3909 tablets (Experimental): Oral administration, 400mg or 600 mg, once a day, and 28 days is a treatment cycle. Continue medication until the disease progresses or intolerant toxicity appears.
  Interventions: Drug: TQB3909 tablet

INTERVENTIONS:
Drug: TQB3909 tablet — TQB3909 is an inhibitor targeting at B-cell lymphoma (BCL)-2 protein.

SUMMARY:
This is a phase Ib/II clinical trial to evaluate the safety and efficacy of TQB3909 tablets in patients with recurrent or refractory CLL/SLL.

ELIGIBILITY:
Inclusion Criteria:

* The subjects volunteered to join the study and signed informed consent form (ICF) with good compliance;
* Age: ≥ 18 years old, ≤75 years old (when signing ICF); Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-1; The expected survival period is more than 3 months;
* Subjects: patients diagnosed as CLL/SLL according to the revised diagnostic criteria of 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines;
* Computed Tomography / Magnetic Resonance Imaging (CT/MRI) of patients with SLL showed measurable lesions;
* Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum pregnancy/urine pregnancy test within 7 days before study enrollment;

Exclusion Criteria:

* Complicated diseases and medical history:

  1. It has appeared or is currently suffering from other malignant tumors within 3 years before the first medication. The following two situations can be included in the group: other malignant tumors treated by single surgery have achieved disease-free survival (DFS) for five consecutive years; Cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  2. Lymphoma/leukemia is known to involve the central nervous system (CNS);
  3. Previously received allogeneic hematopoietic stem cell transplantation;
  4. Received autologous hematopoietic stem cell transplantation within 3 months before the first medication;
  5. Unresolved toxic reaction ≥ CTCAE grade 1 caused by any previous treatment;
  6. Arterial/venous thrombotic events occurred within 6 months before the first medication, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism;
  7. Subjects with any serious and/or uncontrollable diseases;
* Tumor-related symptoms and treatment:

  1. He has received chemotherapy and radiotherapy within 4 weeks before the first medication, immune checkpoint inhibitor and Chimeric Antigen Receptor T (CAR-T)-Cell Immunotherapy within 12 weeks before the first medication, and other small molecule anti-tumor treatments (the elution period is calculated from the end of the last treatment) before the first medication are within 5 half-lives;
  2. previously received BCL-2 inhibitors;
* Research-related treatment: received the vaccine within 4 weeks before the first medication, or planned to be vaccinated during the study;
* Participated in clinical trials of other antineoplastic drugs within 4 weeks before the first medication;
* According to the investigators' judgment, there are patients with accompanying diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who think that there are other reasons that are not suitable for inclusion.
* Allergic to allopurinol and benzbromarone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) | Up to 34 months.
  Incidence of AE evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events 5.0).
Severity of adverse events (AE) | Up to 34 months.
  Severity of AE evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events 5.0).
Incidence of serious adverse events (SAE) | Up to 34 months.
  Incidence of SAE evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events 5.0).
Severity of serious adverse events (SAE) | Up to 34 months.
  Severity of SAE evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events 5.0).
Incidence of abnormal laboratory examination indexes. | Up to 34 months.
  Incidence of abnormal laboratory examination indexes evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events 5.0).
Severity of abnormal laboratory examination indexes. | Up to 34 months.
  Severity of abnormal laboratory examination indexes evaluated by CTCAE 5.0 (Common Terminology Criteria for Adverse Events 5.0).
Recommended phase II dose (RP2D) | Up to 18 months
  To determine the recommended phase II dose of TQB3909 tablets in the treatment of recurrent or refractory CLL/SLL.
Objective remission rate (ORR) determined by Independent Review Committee (IRC) | Up to 34 months
  Determine the objective remission rate (ORR) based on the evaluation results of the Independent Review Committee (IRC), defined as the proportion of subjects whose best remission is complete remission (CR) and partial remission (PR).

SECONDARY OUTCOMES:
Objective remission rate (ORR) determined by the investigators' evaluation. | Up to 34 months
  The objective remission rate (ORR) was determined by the results of the investigator s' evaluation, defined as the proportion of subjects whose best remission is complete remission (CR) and partial remission (PR).
Duration of remission (DOR) | Up to 34 months
  For all subjects whose best response was PR, CR,, the time from the date of first achieving PR, CR to the date of first definite disease progression or death from any cause (whichever occurs first).
Time to disease progression (TTP) | Up to 34 months
  Refers to the time from the first medication to the objective progress of the disease.
Time to remission (TTR) | Up to 34 months
  Time from the beginning of treatment to the first recording of remission (PR or better remission), only the remission population was analyzed.
Progression-free survival (PFS) | Up to 34 months
  The time from the first medication to the objective progression of the disease or death caused from any cause (whichever comes first).
Overall survival (OS) | Up to 34 months
  Time from first dose of study drug to date of death from any cause.
Time to reach maximum concentration (Tmax) | Within 120 hours after administration
  Time to reach maximum plasma concentration after single and multiple dosing of TQB3909 tablets.
Maximum plasma drug concentration (Cmax) | Within 120 hours after administration
  Cmax is the maximum plasma concentration of TQB3909.
Area under the plasma concentration-time curve (AUC0-t) | Within 120 hours after administration
  To characterize the pharmacokinetics of TQB3909 by assessment of area under the plasma concentration time curve.
Plasma elimination half-life (t1/2) | Within 120 hours after administration
  t1/2 is time it takes for the blood concentration of TQB3909 to drop by half.
Undetectable measurable residual disease (U-MRD) ratio of peripheral blood and/or bone marrow. | Up to 34 months
  Refers to the undetected residual lesions. Peripheral blood and/or bone marrow are used to detect less than 1 CLL cell (less than 10-4) in 10000 white blood cells by flow cytometry.
Correlation between potential biomarkers and TQB3909 tablets. | Up to 34 months
  Correlation of potential biomarkers with TQB3909 tablets: such as BTK and PLCG2 mutation status and allele frequency.

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Anqing Municipal Hospital, Anqing, Anhui
  - Gansu province Wuwei tumour hospital, Wuwei, Gansu
  - Sun Yat-Sen University Cancer Canter, Guangzhou, Guangdong
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Harbin first hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Linyi people's hospital, Linyi, Shandong
  - Tai 'an Central Hospital, Tai’an, Shandong
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Peace Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Affiliated hospital of southwest medical university, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang